CLINICAL TRIAL: NCT05779969
Title: Comparison of CT Scan Aspects of the Manubriosternal Joint Between Patients With Axial Spondyloarthritis and Control Subjects
Brief Title: Comparison of CT Scan Between Patients With Axial Spondyloarthritis and Control Subjects
Acronym: SPA-THORAX
Status: Completed | Type: Observational
Sponsor: Hôpital NOVO (Other)
Responsible Party: Sponsor
Other Study IDs: CHRD 2222
Record Dates: First submitted 2023-03-07; First posted 2023-03-22 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Axial Spondyloarthritis
Keywords: Manubriosternal joint,; Axial spondyloarthritis,; Chest CT scan
MeSH Terms: conditions — Axial Spondyloarthritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chest CT scan Patient: Identification of structural damage to the manubriosternal joint (MST) in a population of patients with radiographic axSpA
  Interventions: Other: Chest CT scan
- Chest CT scan Control: Identification of structural damage to the manubriosternal joint (MST) in a control population free of chronic inflammatory rheumatism on chest CT.
  Interventions: Other: Chest CT scan

INTERVENTIONS:
Other: Chest CT scan — Comparison of structural damage to the manubriosternal joint (MST) between a population of patients with radiographic axSpA and a control population free of chronic inflammatory rheumatism on chest CT.

SUMMARY:
The aim of this study is to define structural damage to the manubriosternal joint (MST) in axial spondyloarthritis (axSpA) by comparing its CT scan aspects between a population of patients with radiographic (axSpA) and a control population free of chronic inflammatory rheumatism.

DETAILED DESCRIPTION:
Axial spondyloarthritis (axSpA) is, together with rheumatoid arthritis, one of the 2 major chronic inflammatory rheumatic diseases. While the lumbar spine and sacroiliac joints are at the forefront of the clinic and diagnosis of axSpA, clinical involvement of the rib cage is common and long-standing. It can lead to limitation of thoracic extension and respiratory consequences. Clinical involvement of the anterior chest wall was evaluated in the early 2010s in axSpA, especially in the newer forms.

Several anatomical structures of the thoracic cage can be the cause of pain and among these is the manubriosternal joint (MST). It is known to be a possible site of inflammatory involvement in axSpA and this is well demonstrated by MRI imaging. Bone CT scans allow precise analysis of changes in the MST joint, but unlike MRI, they do not analyse inflammation, which is itself the cause of structural changes. While inflammation is the main cause of pain, structural changes, particularly ankylosis, are the cause of potentially disabling sequelae. To date, there have been no studies of structural damage to the MST joint in patients with axSpA, including the radiographic form. Moreover, little is known about the CT scan data of the MST joint in healthy subjects. Apart from the interest in defining axSpA-related abnormalities for CT scan analysis of the MST joint in general, it is important to know the frequency and types of structural abnormalities of the MST joint in axSpA, not for early diagnosis, but in terms of assessing the severity of the disease.

The investigator's hypothesis is that there are structural abnormalities of the STD joint in the radiographic axSpA, the characteristics, prevalence and relationship to patient and disease characteristics of which must be determined. This should be analysed in the non-radiographic axSpA. This requires comparison with a control population, but as there are no validated criteria for assessing the pathological nature of the STD joint on CT, it is necessary to proceed in 2 steps:

1. - To define the structural damage to the MST joint in radiographic axSpA by comparison with control subjects. This comparison should focus first on the various basic abnormalities known to be present in radiographic axSpA, and in particular in the sacroiliac joints, such as erosions, subchondral bone condensation, pinching of the joint space, and ankylosis, which should be compared to the fusion phenomena described in controls.
2. - Study the characteristics of this structural damage in radiographic and non-radiographic axSpA.

ELIGIBILITY:
Inclusion Criteria :

axSpA population:

* Adults aged 18 to 69 years,
* Diagnosis of axSpA according to the ASAS 2009 criteria,
* Hospitalized in the Rheumatology Department of the NOVO Hospital (Pontoise site) from 01/01/2015 to 30/10/2022 and had a Chest CT scan with images available in the hospital's computer system,
* Informed of the study and did not object.

Control population:

* Adults aged 18 to 69 years,
* Day hospitalization in the pneumology department of the NOVO Hospital (Pontoise site) from 01/01/2015 to 30/10/2022 and having had a lung scan on this occasion,
* Informed of the study and did not object.

Exclusion Criteria :

axSpA population:

* Peripheral spondyloarthritis,
* Unavailability of chest CT scan images in the hospital computer system,
* Unknown result of pelvic X-ray.

Control population:

* Lung cancer or suspected lung cancer
* Any of the following conditions: spondyloarthritis, rheumatoid arthritis, psoriatic arthritis, SAPHO syndrome, chest wall bone disease, tumour bone disease, severe scoliosis, malformative syndrome
* History of thoracic trauma or thoracic surgery,
* Unavailability of chest CT scan images in the hospital computer system.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients having a Chest CT scan (as part of a conventional hospitalization or Day hospitalization) between 01/01/2015 and 30/10/2022 for a population of patients with radiographic axSpA and a control population free of chronic inflammatory rheumatism
Sampling Method: Non-Probability Sample
Enrollment: 377 (Actual)
Dates: Start 2023-02-09 (Actual); Primary Completion 2024-12-13 (Actual); Study Completion 2024-12-13 (Actual)

PRIMARY OUTCOMES:
To define the structural damage of the manubriosternal joint (MST) in axSpA by comparing its Chest CT scan aspects between a population of patients with radiographic axSpA and a control population free of chronic inflammatory rheumatism | At the end of the study, an average of 1 month
  Assessment of the various aspects of the manubriosternal joint on the CT scan. These different elements of analysis are grouped in an evaluation grid. Assessment of the various aspects of the manubriosternal joint on the CT scan. These different elements of analysis are grouped in an evaluation grid. The prevalence of each unit anomaly (e.g. "erosions") will be compared between the radiographic axSpA population and the control population.

SECONDARY OUTCOMES:
Determination of the prevalence of structural damage to the manubriosternal joint (MST) in radiographic axSpA by comparing this population with the control population | At the end of the study, an average of 1 month
  Structural damage to the manubriosternal joint will be assessed on the scans by a double radiologist/rheumatologist reading in the different populations using a review grid.
Determination of the prevalence of structural damage to the manubriosternal joint (MST) in non-radiographic axSpA by comparing this population with the control population | At the end of the study, an average of 1 month
  Structural damage to the manubriosternal joint will be assessed on the scans by a double radiologist/rheumatologist reading in the different populations using a review grid.
Determination of the prevalence of structural damage to the manubriosternal joint (MST) between radiographic axSpA and non- radiographic axSpA | At the end of the study, an average of 1 month
  Structural damage to the manubriosternal joint will be assessed on the scans by a double radiologist/rheumatologist reading in the different populations using a review grid.
Search for a significant association between a phenotypic feature of axSpA and the existence of structural damage to the manubriosternal joint (MST) | At the end of the study, an average of 1 month
  The phenotypic character of axSpA is assessed by clinical criteria defined by the rheumatologist

CONTACTS AND LOCATIONS:
Overall Officials: Dr Edouart Pertuiset, Principal Investigator — Hospital NOVO - Pontoise site
Locations (1):
- Rheumatology department - NOVO Hospital - Pontoise site, Pontoise, France

REFERENCES:
- [Background] Taurog JD, Chhabra A, Colbert RA. Ankylosing Spondylitis and Axial Spondyloarthritis. N Engl J Med. 2016 Jun 30;374(26):2563-74. doi: 10.1056/NEJMra1406182. No abstract available. PMID 27355535
- [Background] van der Linden S, Valkenburg HA, Cats A. Evaluation of diagnostic criteria for ankylosing spondylitis. A proposal for modification of the New York criteria. Arthritis Rheum. 1984 Apr;27(4):361-8. doi: 10.1002/art.1780270401. PMID 6231933
- [Background] Rudwaleit M, van der Heijde D, Landewe R, Listing J, Akkoc N, Brandt J, Braun J, Chou CT, Collantes-Estevez E, Dougados M, Huang F, Gu J, Khan MA, Kirazli Y, Maksymowych WP, Mielants H, Sorensen IJ, Ozgocmen S, Roussou E, Valle-Onate R, Weber U, Wei J, Sieper J. The development of Assessment of SpondyloArthritis international Society classification criteria for axial spondyloarthritis (part II): validation and final selection. Ann Rheum Dis. 2009 Jun;68(6):777-83. doi: 10.1136/ard.2009.108233. Epub 2009 Mar 17. PMID 19297344
- [Background] Elhai M, Paternotte S, Burki V, Durnez A, Fabreguet I, Koumakis E, Meyer M, Payet J, Roure F, Dougados M, Gossec L. Clinical characteristics of anterior chest wall pain in spondyloarthritis: an analysis of 275 patients. Joint Bone Spine. 2012 Oct;79(5):476-81. doi: 10.1016/j.jbspin.2011.10.003. Epub 2011 Nov 25. PMID 22119315
- [Background] Wendling D, Prati C, Demattei C, Loeuille D, Richette P, Dougados M. Anterior chest wall pain in recent inflammatory back pain suggestive of spondyloarthritis. data from the DESIR cohort. J Rheumatol. 2013 Jul;40(7):1148-52. doi: 10.3899/jrheum.121460. Epub 2013 May 15. PMID 23678156
- [Background] Weber U, Lambert RG, Rufibach K, Maksymowych WP, Hodler J, Zejden A, Duewell S, Kissling RO, Filipow PL, Jurik AG. Anterior chest wall inflammation by whole-body magnetic resonance imaging in patients with spondyloarthritis: lack of association between clinical and imaging findings in a cross-sectional study. Arthritis Res Ther. 2012 Jan 6;14(1):R3. doi: 10.1186/ar3551. PMID 22226453
- [Background] Cameron HU, Fornasier VL. The manubriosternal joint--ananatomicoradiological survey. Thorax. 1974 Jul;29(4):472-4. doi: 10.1136/thx.29.4.472. PMID 4854943